CLINICAL TRIAL: NCT07238075
Title: A First-in-human, Multicenter Dose Escalation and Multiple Cohort Expansion Phase 1a/b Study to Investigate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ADCX-020 in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: ADCX-020 for the Treatment of Patients With Locally Advanced or Metastatic Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adcytherix SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCX-020-01; 2025-523959-65-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignancy; Advanced Solid Cancers; Metastatic Solid Tumors
Keywords: Antibody Drug Conjugate; Antineoplastic Agents; Monoclonal Antibodies; Neoplasms; Response Evaluation Criteria in Solid Tumors (RECIST); Phase 1 clinical trial; Maximum Tolerated Dose; Open-Label Trials; Multicenter Study; Pharmacokinetics; Pharmacodynamics; Drug-Related Side Effects and Adverse Reactions; Dose-Response Relationship, Drug; Adults; Progression-Free Survival / Overall Survival; Overall response rate
MeSH Terms: conditions — Neoplasms; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a ADCX-020 (Experimental): Dose escalation of ADCX-020, intravenous
  Interventions: Drug: ADCX-020
- Phase 1b: ADCX-020 (Experimental): Dose optimization and expansion of ADCX-020, intravenous
  Interventions: Drug: ADCX-020

INTERVENTIONS:
Drug: ADCX-020 — ADC

SUMMARY:
The purpose of this first-in-human study is to explore the safety, pharmacokinetics and effects of the study drug ADCX-020 in patients with advanced and metastatic solid tumors. ADCX-020 is an investigational anticancer therapy called antibody drug conjugate.

This study is set up in multiple parts. In the first part of the study, participants receive increasing doses of ADCX-020. Then 2 or more doses will be assessed to identify the optimal dose. This optimal dose is subsequently evaluated for effect on different cancer types.

DETAILED DESCRIPTION:
This is a first-in-human (FIH) open-label, multicenter, dose escalation and multiple cohort expansion Phase 1a/b study to investigate safety, tolerability, PK, pharmacodynamics, and preliminary efficacy of ADCX-020 monotherapy in participants with relapsed or refractory solid tumors, or who are intolerant to standard of care.

During dose escalation, Phase 1a, participants will receive escalating doses of ADCX-020 to identify the MTD based on the observation of DLTs. Intermediate and higher dose levels as well as alternative dosing regimens may be investigated during this part of the study.

Dose expansion, Phase 1b, will be initiated with a dose optimization of ADCX-020 using two or more dose levels of ADCX-020 and/or evaluating a different dosing regimen. Expansion in multiple cohorts is planned for selected patient populations using the RP2D.

Phase 1a will be overseen by a Dose Escalation Committee (DEC) and Phase 1b will be overseen by a Safety Review Committee (SRC).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years of age
* Ph1a: Locally advanced or metastatic solid tumor relapsed or PD following local standard treatments, for which no standard treatment is available
* Ph1b: Eligible patients should have only received prior lines of systemic therapy according to SoC in the advanced/metastatic setting (not counting neoadjuvant/adjuvant treatment if completed >6 months prior to recurrence)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Radiologically measurable disease by RECIST v1.1
* Mandatory adequate tumor tissue sample available
* Must have recovered from all clinically relevant toxicities from previous cancer therapies (to at least Grade 1, except for alopecia)

Exclusion Criteria:

* Known allergies/hypersensitivity/intolerance to or contraindication to exatecan, or any excipient
* Phase 1b: Prior antibody drug conjugate exposure with a topoisomerase 1 inhibitor payload
* Uncontrolled or significant cardiac disease including left ventricular ejection fraction (LVEF) <50%, myocardial infarction or uncontrolled/unstable angina
* Has clinically active central nervous system (CNS) metastases
* Has a history of lung fibrosis or non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Active corneal disease, or history of corneal disease within 12 months prior to enrollment
* Other unacceptable abnormalities, medications or procedures as defined by protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Ph1a: To determine the safety and tolerability of ADCX-020 | Start of treatment until 30 days after last dose
  Incidence and severity of treatment-emergent adverse events (TEAEs)
Ph1a: To determine the maximun tolerated dose (MTD) or recommended dose range for expansion and optimization | Start of treatment to end of DLT observation period
  Incidence of dose-limiting toxicities (DLTs) at different dose levels
Ph1b: To determine the recommended Phase 2 dose (RP2D) | Baseline to 30 days post last study drug administration
  Cumulative incidence and severity of TEAEs, preliminary anti-tumor activity and pharmacokinetics and -dynamics findings
Ph1b: To assess the objective response rate (ORR) of ADCX-020 | Baseline until the date of the first documented disease progression, death, or start of new anticancer therapy (approximately 24 months)
  Preliminary efficacy based on ORR assessed by Investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
To evaluate duration of objective response (DoR) | Baseline until approximately 24 months
  DoR is defined as the time from first documented response to the date of first PD or death due to any cause
To evaluate the disease control rate (DCR) | Baseline until approximately 24 months
  DCR is defined as the proportion of participants who achieved an objective response or stable disease, per RECIST v1.1.
To assess prgression free survival (PFS) | Baseline until approximately 24 months
  PFS is defined as the time from first dose date to the date of first documented disease progression per RECIST v1.1 or death due to any cause
Phase 1b: To evaluate overall survival (OS) | Baseline to approximately 24 months
  OS as time from study start to the date of death due to any cause
To determine the plasma concentration of ADCX-020 | Start of treatment until 30 days after last dose
  PK analysis for Cmax and Cmin
To determine the time to Cmax (Tmax) for ADCX-020 | Start of treatment until 30 days after last dose
  PK analysis for Tmax
To determine the terminal phase elimination half-life (t1/2) for ADCX-020 | Start of treatment until 30 days after last dose
  PK analysis for t1/2
To determine the area under the plasma concentration-time curve (AUC) for ADCX-020 | Start of treatment until 30 days after last dose
  PK analysis for AUC
To evaluate the immunogenicity of ADCX-020 | Start of treatment until 30 days after last dose
  Frequency of participants developing anti-ADCX-020 antibodies and titer assessments

CONTACTS AND LOCATIONS:
Overall Officials: Adcytherix, Study Director — Adcytherix SAS

IPD SHARING:
Plan to Share IPD: No